CLINICAL TRIAL: NCT00840918
Title: The Effect of Perioperative Intravenous Lidocaine on Postoperative Outcomes After Cardiac Surgery
Brief Title: Intravenous Lidocaine and Postoperative Outcomes After Cardiac Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Problem with enrollment
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 08-861
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Atrial Fibrillation
Keywords: Cardiac surgery; Lidocaine; Quality of life
MeSH Terms: conditions — Atrial Fibrillation | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Intravenous Lidocaine group
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): Intravenous placebo Group - Placebo is administered intravenously throughout surgery and during the 24 hours following surgery
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lidocaine — Intravenous Lidocaine Group - Lidocaine administered intravenously throughout surgery and during the 24 hours following surgery.
  Arms: 1
Other: Placebo — Placebo is administered intravenously throughout surgery and during the 24 hours following surgery
  Arms: Placebo

SUMMARY:
This study is being done to determine if lidocaine, administered during surgery and for 24 hours after surgery can reduce inflammation, thereby reducing the risk of atrial fibrillation and 30 day mortality after surgery. Participants undergoing cardiac surgery will be randomized to receive either lidocaine or placebo.

DETAILED DESCRIPTION:
Subjects undergoing cardiac surgery are randomized into one of two groups.

* Group 1: Intravenous Lidocaine Group
* Group 2: Intravenous placebo Group

Either Lidocaine or placebo is administered throughout surgery and 24 hours after surgery.

Patients in both groups will undergo quality of life assessments and functional recovery assessments post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90 years old
* Scheduled for cardiac surgery requiring cardiopulmonary bypass
* Written informed consent

Exclusion Criteria:

* Off-pump surgical procedures
* Anticipated deep hypothermic circulatory arrest
* Any contraindications to the proposed interventions including lidocaine allergy
* History of preoperative atrial fibrillation
* Baseline Screening revealing preexisting dementia or delirium
* Preoperative liver failure defined as Child-Pugh Score > 6

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2009-02; Primary Completion 2014-12-15 (Actual); Study Completion 2014-12-15 (Actual)

PRIMARY OUTCOMES:
atrial fibrillation | postoperatively
  To test the hypothesis that lidocaine infusion started at induction of anesthesia and maintained for 24 hours postoperatively will decrease the incidence of atrial fibrillation compared to an intravenous saline control.
mortality | 30 days post surgery
  To test the hypothesis that lidocaine infusion started at induction of anesthesia and maintained for 24 hours postoperatively will decrease the incidence of 30 day mortality as compared to an intravenous saline control.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Grady, M.D., Principal Investigator — The Cleveland Clinic; Daniel I Sessler, M.D., Study Chair — The Cleveland Clinic
Locations (1):
- SAL Hospital, Ahmedabad, Gujarat, India